CLINICAL TRIAL: NCT06793319
Title: Atriyal Fibrilasyonu Olan Hastalara Verilen Eğitimin Anksiyete Düzeyleri Üzerine Etkisi
Brief Title: The Effect of Education Given to Patients with Atrial Fibrillation on Anxiety Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kübra Kocaispir (Other)
Responsible Party: Sponsor-Investigator, Kübra Kocaispir, Intensive Care Nurse, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 61351342/020-192
Record Dates: First submitted 2024-12-28; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation New Onset
Keywords: Anxiety; Atrial Fibrillation; Patient education
MeSH Terms: conditions — Atrial Fibrillation; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: It is a study that does not involve drugs or biological products. It was examined how the education given to patients affected anxiety. The operating model is parallel.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- training group (Experimental): Written and verbal consent of the training group patients was obtained using the Patient Information and Consent Form. The patients in the training group first filled out the Personal Information Form and Situationality Anxiety Inventory (STAI 1) before the training. Atrial Fibrillation training was given one-on-one in the patient's room. The training was explained using clear, simple language that patients could understand. Patients were encouraged to ask questions. They were asked about the parts they did not understand. It was done by answering the patients' questions. The training was held in 2 sessions in one day. It was planned as one hour before noon and one hour in the afternoon. After the Atrial Fibrillation training given to the patients, the Situationality Anxiety Inventory (STAI 1) was filled out again to evaluate the anxiety level.
  Interventions: Other: educational app
- control group (No Intervention): Written and verbal consent of the patients in the control group was obtained using the Patient Information and Consent Form. Personal Information Form and Situationality Anxiety Inventory (STAI 1) were filled out. No training was given. At the end of the follow-up period, the Situationality Anxiety Inventory (STAI 1) was filled out again.

INTERVENTIONS:
Other: educational app — State Anxiety Inventory was filled out before the training. Atrial Fibrillation training was provided. After the training, the Situationality Anxiety Inventory was filled out again. It was aimed to evaluate the effect of education on anxiety.
  Arms: training group

SUMMARY:
This study aims to evaluate the effect of a structured training program on state anxiety levels in patients diagnosed with Atrial Fibrillation (AF). AF is a chronic heart rhythm disorder that negatively affects patients' quality of life with both physical and psychological symptoms. Lack of information and uncertainty in AF patients cause increased anxiety levels, making compliance with treatment difficult. This study aims to determine whether an educational intervention for AF patients can reduce their anxiety levels and increase their awareness of the disease. This is a randomized controlled trial. A two-session individual training program containing detailed information about AF will be applied to the training group and no training will be given to the control group. Data will be collected through a personal information form and the Situationality Anxiety Inventory (STAI).

Hypotheses of the Research H0: Training regarding Atrial Fibrillation has no effect on the anxiety level of patients.

H1: Education regarding Atrial Fibrillation reduces the anxiety level of patients.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed with AF,
* Able to speak and understand Turkish,
* Does not have a physical or psychological disorder that would cause communication problems,
* Patients between the ages of 18 and 65 who are oriented to place and time, -Agreeing to participate in the study

Exclusion criteria:

* Using any psychotropic medication (antidepressant, anxiolytic, antipsychotic)

Ages: 18 Months to 65 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Anxiety Levels of Patients Given Atrial Fibrillation Training | Within 2-3 hours after training
  This study was conducted in a randomized controlled manner. It was done with 60 patients. 30 patients were assigned to the training group and 30 patients to the control group. There is a training and control group. Groups will fill out a personal information form and the State Anxiety Inventory. Atrial fibrillation training was given to the training group and the state anxiety inventory (STAI 1) was filled out again. The control group was not given any training and had a state anxiety inventory filled out. The data obtained in the study were analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Number, percentage, mean and standard deviation were used as descriptive statistical methods in the evaluation of the data. Differences between the proportions of categorical variables in independent groups were analyzed with Chi-Square tests. Kurtosis and Skewness values were examined to determine whether the research variables showed normal distribution

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat B Ateş, Study Director — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPDs can result in a broadcast
Supporting Information: Study Protocol, SAP, ICF, CSR